CLINICAL TRIAL: NCT05577962
Title: The Effect of Opioid-free Anesthesia Protocol on the Early Quality of Recovery After Thyroidectomy (TOFA Trial): Study Protocol for a Prospective, Monocentric, Randomized, Single-blinded Trial
Brief Title: Opioid Free Anesthesia on the Quality of Early Recovery
Acronym: opioid-free
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: opioid-free anesthesia
Record Dates: First submitted 2022-10-07; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Opioid-free Anesthesia
Keywords: thyroidectomy; the early quality of recovery
MeSH Terms: interventions — Sensitivity Training Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C group (No Intervention): The routine anesthesia group
- T group (Experimental): Opioid-free Anesthesia
  Interventions: Drug: T group

INTERVENTIONS:
Drug: T group — OFA scheme (group T) was given dexamethasone 8mg for anti-inflammatory and antiemetic before operation, flurbiprofen axetil 50mg for preemptive analgesia, and dexmedetomidine was infused under ECG monitoring at an initial rate of 0.5 μ G/kg (more than 10min), then changed to 0.2ug/kg/h, and stopped infusion 20 minutes before operation closure. Before induction, lidocaine (1mg/kg), esketamine (0.5mg/kg), propofol (1-2mg/kg) and rocuronium (0.6mg/kg) were infused slowly, and endotracheal intubation was carried out when the anesthetic was fully effective and the BIS value was about 40. After successful intubation, an experienced anesthesiologist guided by ultrasound performed bilateral superficial cervical plexus block with 0.5% ropivacaine and injected 3-4ml at two points respectively; During the operation, sevoflurane (MAC1.0 - 1.4) was used to maintain the depth of anesthesia
  Arms: T group

SUMMARY:
To analyze and compare the effect of OFA scheme and traditional balanced anesthesia scheme on QoR15 after thyroidectomy, and further clarify the safety and rationality of OFA scheme in perioperative application of thyroid surgery.

DETAILED DESCRIPTION:
OFA scheme (group T) was given dexamethasone 8mg for anti-inflammatory and antiemetic before operation, flurbiprofen axetil 50mg for preemptive analgesia, and dexmedetomidine was infused under ECG monitoring at an initial rate of 0.5 μ G/kg (more than 10min), then changed to 0.2ug/kg/h, and stopped infusion 20 minutes before operation closure. Before induction, lidocaine (1mg/kg), esketamine (0.5mg/kg), propofol (1-2mg/kg) and rocuronium (0.6mg/kg) were infused slowly, and endotracheal intubation was carried out when the anesthetic was fully effective and the BIS value was about 40. After successful intubation, an experienced anesthesiologist guided by ultrasound performed bilateral superficial cervical plexus block with 0.5% ropivacaine and injected 3-4ml at two points respectively; During the operation, sevoflurane (MAC1.0 - 1.4) was used to maintain the depth of anesthesia; The routine anesthesia group (Group C) was induced to give sufentanil 0.3-0.5ug/kg, propofol 1-2mg/kg, rocuronium 0.6mg/kg slowly, and then intubated when the anesthetic was fully effective and the BIS value was about 40. Remifentanil was continuously pumped 0.1-0.2ug/kg during operation min； Combined with sevoflurane (MAC 0.8-1) to maintain the depth of anesthesia.

ELIGIBILITY:
Inclusion Criteria

* Patients undergoing elective thyroidectomy under general anesthesia
* >18 year old
* The informed consent form has been signed
* American Society of Anesthesiologists (ASA) anesthesia grade I - II

Exclusion Criteria:

* Long term use of opioids
* Long term use of NSAIDs
* Have a history of psychosis, epilepsy, preoperative anxiety, depression, and emotional management disorders
* Patients with increased gastric contents reflux and respiratory tract aspiration
* Operation time>3h
* Severe liver and kidney insufficiency, cardiac insufficiency, bradycardia with 2 ° II or 3° atrioventricular block
* Those who are allergic to or have contraindications to drugs that may be used in the test
* Those who cannot cooperate with researchers

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 160 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The QoR-15 score | Hour 24，Hour 48，Hour 72 after surgery
  The quality of recovery-15 score,The QoR was classified as excellent (QoR-15 > 135), good (122 ≤ QoR-15 ≤ 135), moderate (90 ≤ QoR-15 ≤ 121) or poor (QoR-15 < 90).

SECONDARY OUTCOMES:
Postoperative VAS score | Hour 24，Hour 48，Hour 72 after surgery
  Postoperative Visual Analog Scale score, For measurement of the magnitude of pain, the most used scale is "no pain" (corresponding to the scale of 0) and "pain too intense to be tolerated" (corresponding to the scale of 100)
Postoperative complication rate | Hour 24，Hour 48，Hour 72 after surgery
  Postoperative complication rate
Opioid consumption | Hour 24，Hour 48，Hour 72 after surgery
  morphine or equivalent daily consumption after surgery if necesssary
Anesthesia related adverse events | Hour 24，Hour 48，Hour 72 after surgery
  Anesthesia related adverse events
Postoperative fatigue, ICFS scores after surgery | Hour 24，Hour 48，Hour 72 after surgery
  Identity-Consequence Fatigue Scale (ICFS) in patients was used to assess the intensity of fatigue.A questionnaire was developed using the 48 items that remained following the content analysis. All items were rated on six-point adjectival scales with anchors from "not at all" to "all of the time" or "not at all" to "more often than usual."
Postoperative mental state | Hour 24，Hour 48，Hour 72 after surgery
  Postoperative Mini-Mental State Examination (MMSE) scores.MMSE <27 was taken to indicate cognitive impairment.
Incidence of chronic pain and quality of life | 3 months after surgery
  Incidence of chronic pain and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Haijun Hou, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Haijun Hou, Beijing, China

IPD SHARING:
Plan to Share IPD: No